CLINICAL TRIAL: NCT00709397
Title: HIV-1 Viral Dynamics in Subjects Initiating Raltegravir Therapy
Status: Terminated | Type: Observational
Why Stopped: lack of accrual
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Daniel R. Kuritzkes, MD, Brigham and Women's Hospital
Other Study IDs: 2007-P-002410/1
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Last update posted 2010-08-02 (Estimated); Status verified 2010-07

CONDITIONS: HIV-1 Infection
Keywords: HIV-1; drug resistance; raltegravir; integrase inhibitor
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood mononuclear cells will be tested for HIV-1 DNA levels. The cell pellets obtained from each of the samples will be tested for 1) total HIV-1 DNA and 2-LTR circles using real-time quantitative PCR and 2) integrated proviral DNA using Alu real-time nested PCR.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation: antiretroviral-experienced patients requiring raltegravir to construct an adequately potent antiretroviral regimen.
  Interventions: Other: blood drawing

INTERVENTIONS:
Other: blood drawing — Subjects will have been prescribed raltegravir (400 mg BID) by their primary physicians. Such subjects will have frequent blood sampling in this study to monitor the virologic response to raltegravir therapy.

SUMMARY:
This study is designed to determine how quickly HIV-1 is cleared from the blood in treatment-experienced patients beginning a salvage therapy regimen that includes the integrase inhibitor raltegravir. The hypothesis is that HIV-1 is cleared as rapidly in these patients as in treatment-naive patients starting a raltegravir-based regimen.

DETAILED DESCRIPTION:
This pilot study will closely examine the viral dynamics of both HIV-1 RNA and DNA in treatment-experienced subjects initiating raltegravir. The data derived from this study will further elucidate the effects of antiviral therapy on viral decay and help refine current viral dynamics models. In addition, results of this study will generate hypotheses for further testing regarding the mechanisms of action of integrase inhibitor therapy in salvage regimens. Lastly, this viral dynamic study on a unique cohort will provide an opportunity to further validate the effectiveness of the methods of measuring rate of decrease of viral RNA and DNA in piloting potential potent drug regimens.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected patients age 18 years or older requiring treatment with raltegravir in order to construct an adequately active antiretroviral regimen.
* Availability of at least two other drugs expected to have full activity based on genotypic and/or phenotypic drug resistance testing, a co-receptor tropism assay, or first use of a drug from a previously unused class of antiretroviral drugs (e.g., first use of enfuvirtide).
* Plasma HIV-1 RNA >10,000 copies/mL at screening (within 6 weeks of study entry).
* Negative serum or urine pregnancy test at screening and within 48 hours prior to entry for women with reproductive potential
* Ability and willingness of subject or legal guardian/representative to provide informed consent.

Exclusion Criteria:

* Pregnancy or breast-feeding.
* Previous treatment with any approved or investigational strand-transfer integrase inhibitor at any time prior to study entry.
* Known allergy/sensitivity or any hypersensitivity to components of study drugs or their formulation.
* Any subject with an acute AIDS-defining opportunistic infection (OI) who is not clinically stable or who has not been on therapy for the OI for at least 30 days prior to study entry. Subjects who have no evidence of active disease and are receiving maintenance therapy for AIDS-related OIs will be eligible.
* Treatment within 30 days prior to study entry with immune modulators such as systemic steroids, interleukins, interferons, granulocyte colony-stimulating factor (G-CSF), erythropoietin, or any investigational therapy.

NOTE: Subjects receiving stable physiologic glucocorticoid doses, defined as prednisone ≤ 10 mg/day (or equivalent) as a stable or tapering dose, will be permitted. Subjects receiving corticosteroids for acute therapy forPneumocystis jaroveci pneumonia (PCP) or asthma exacerbation, or receiving a short course (defined as ≤ 2 weeks of pharmacologic glucocorticoid therapy) will not be excluded.

• Serious illness requiring systemic treatment and/or hospitalization until candidate either completes therapy or is clinically stable on therapy, in the opinion of the site investigator, for at least 7 days prior to study entry.

NOTE: Oral candidiasis, vaginal candidiasis, mucocutaneous herpes simplex, and other minor illnesses (as judged by the site investigator) have no restriction.

• Substance abuse that, in the opinion of the site investigator, would interfere with adherence to study requirements.who have limited or no treatment options due to extensive antiretroviral drug resistance or drug intolerance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible subjects are antiretroviral-experienced patients requiring raltegravir to construct an adequately potent antiretroviral regimen.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2008-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
first- and second-phase decay rates of plasma HIV-1 RNA | 24 weeks

SECONDARY OUTCOMES:
1. As exploratory analyses, to compare the observed first-phase decay rate of plasma HIV-1 RNA in treatment-experienced patients receiving raltegravir to treatment-naïve patients in other studies. | 24 weeks
2. Quantify changes in the intracellular levels of HIV-1 proviral DNA and LTR circles during raltegravir therapy. | 24 weeks
3. Correlate changes in the intracellular DNA compartments with first- and second-phase plasma HIV-1 RNA clearance rates. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Daniel R Kuritzkes, MD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts